CLINICAL TRIAL: NCT04232345
Title: A Phase I, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD4831 Following Multiple-ascending Dose Administration in Japanese and Chinese Healthy Volunteers
Brief Title: A Study to Assess the Effect AZD4831 in Japanese and Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D6580C00008
Record Dates: First submitted 2020-01-03; First posted 2020-01-18 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)
Keywords: Randomized; Single-blind; Placebo-controlled; Multiple-ascending dose; AZD4831 oral suspension
MeSH Terms: interventions — AZD4831

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, single-blind, placebo-controlled, MAD sequential-group study in healthy Japanese (Part 1, Cohorts 1, 2, and 3) and Chinese (Part 2, Cohort 4) male subjects, conducted at a single study center. Up to 40 healthy male subjects aged 18 to 50 years (inclusive) are planned to be investigated in 4 cohorts, but up to 5 cohorts may be included if the SRC considers it necessary to repeat a dose level or if additional dose levels are required.
  Up to 8 subjects will participate in each cohort. Within each cohort 6 subjects will be randomly assigned to receive AZD4831 and 2 subjects to receive placebo. AZD4831 or placebo will be administered once daily for a period of 10 days. It is anticipated this will be sufficient to achieve and maintain steady state pharmacokinetic (PK) profiles for several days, permitting evaluation of the safety and tolerability of multiple dose. The subjects will stay at the study center during the whole dosing period and until 48 hours.
Who Masked: Participant
Masking Description: This study is single-blind with regards to treatment (AZD4831 or placebo) at each dose level. AZD4831 and placebo will be matched for appearance and amount. Subjects randomized to placebo will receive the same volume of oral suspension as subjects on active drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Part 1): AZD4831 Dose 1 (Experimental): Randomized subjects will receive oral suspension of AZD4831 Dose 1 once daily in the morning for a period of 10 days
  Interventions: Drug: AZD4831
- Cohort 2 (Part 1): AZD4831 Dose 2 (Experimental): Randomized subjects will receive oral suspension of AZD4831 Dose 2 once daily in the morning for a period of 10 days.
  Interventions: Drug: AZD4831
- Cohort 3 (Part 1): AZD4831 Dose 3 (Experimental): Randomized subjects will receive oral suspension of AZD4831 Dose 3 once daily in the morning for a period of 10 days.
  Interventions: Drug: AZD4831
- Cohort 4 (Part 2): AZD4831 Dose 2 (Experimental): Randomized subjects will receive oral suspension of AZD4831 Dose 2 once daily in the morning for a period of 10 days.
  Interventions: Drug: AZD4831
- Placebo (Part 1) (Experimental): Randomized subjects will receive oral suspension of placebo once daily in the morning for a period of 10 days.
  Interventions: Drug: Placebo
- Placebo (Part 2) (Experimental): Randomized subjects will receive oral suspension of placebo once daily in the morning for a period of 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4831 — Subjects will be fasted for at least 10 hours before receiving the AZD4831 in the form of an oral suspension.
  Arms: Cohort 1 (Part 1): AZD4831 Dose 1; Cohort 2 (Part 1): AZD4831 Dose 2; Cohort 3 (Part 1): AZD4831 Dose 3; Cohort 4 (Part 2): AZD4831 Dose 2
Drug: Placebo — Subjects will be fasted for at least 10 hours before receiving the placebo in the form of an oral suspension.
  Arms: Placebo (Part 1); Placebo (Part 2)

SUMMARY:
This study is randomized, single-blind, placebo-controlled Phase 1 study aimed to assess the safety and efficacy, pharmacokinetics and pharmacodynamics of multiple doses of oral AZD4831 in healthy Japanese and Chinese volunteers

DETAILED DESCRIPTION:
This is a Phase I, randomized, single-blind, placebo-controlled, multiple-ascending dose (MAD), sequential-group study in healthy Japanese (Part 1, Cohorts 1, 2, and 3) and Chinese (Part 2, Cohort 4) male subjects, conducted at a single study center. Four cohorts are planned, but one additional cohort may be enrolled based on a Safety Review Committee (SRC) decision.

The 4 multiple dose levels are planned as follows:

* Cohort 1: Dose 1
* Cohort 2: Dose 2
* Cohort 3: Dose 3
* Cohort 4: Dose 2

A randomization ratio of 3:1 (AZD4831 versus placebo) will be used.

For each cohort the study will comprise:

* Screening Period of a maximum of 28 days.
* A Treatment Period during which subjects are resident in the study center from the day before first dosing with the Investigational Medicinal Product (Day -1) until at least 48 hours after last dosing on Day 10; subjects will be discharged on Day 12.
* Three Follow-up Visits on Day 14, Day 16 (±1 day), and Day 20 (±1 day).
* A Final Follow-up Visit on Day 24 (±2 days).

Each subject will be involved in the study for 8 to 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male Japanese and Chinese subjects aged 18 - 50 years (inclusive at Screening) with suitable veins for cannulation or repeated venipuncture.

A Japanese subject is defined as having both parents and 4 grandparents who are ethnically Japanese. This includes second and third generation Japanese whose parents or grandparents are living in a country other than Japan.

A Chinese subject is defined as having both parents and 4 grandparents who are ethnically Chinese. This includes second and third generation Chinese whose parents or grandparents are living in a country other than China.

* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Provision of signed, written and dated informed consent for optional genetic/biomarker research. If a subject decline to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this protocol.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Presence of infection(s) (particularly fungal infection), as judged by the Investigator.
* History of, or current thyroid disease.
* Any ongoing skin disorder, history of or ongoing clinically significant allergy/hypersensitivity.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the Investigator at Screening and/or Day -1.

  1. Alanine transaminase (ALT) not within normal range
  2. Aspartate aminotransferase (AST) not within normal range
  3. Creatinine not within normal range
  4. White blood cell (WBC) count not within normal range
  5. Hemoglobin not within normal range;
  6. Estimated Glomerular Filtration Rate (eGFR) not within normal range.
* Any positive result at Screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV) type 1 and 2.
* Abnormal vital signs, after 10 minutes supine rest, at Screening and/or Day -1, defined as any of the following:

  1. SBP < 90 mmHg or ≥ 140 mmHg.
  2. DBP < 50 mmHg or ≥ 90 mmHg.
  3. Pulse < 45 or > 85 bpm.
* Any clinically significant abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and/or any clinically significant abnormalities in the 12-lead ECG, as judged by the Investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy at Screening and/or Day -1.
* Prolonged QTcF > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome at Screening and/or Day -1.
* PR(PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation) at Screening and/or Day -1.
* PR(PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third-degree atrioventricular (AV)-block, or AV dissociation at Screening and/or Day -1.
* Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or interventricular conduction delay with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of, for example, ventricular hypertrophy or pre-excitation at Screening and/or Day -1.
* Electrocardiogram findings suggesting a metabolic or other non-cardiac condition that may confound interpretation of serial changes (such as hypokalemia) at Screening and/or Day -1.
* Known or suspected history of drug abuse as judged by the Investigator.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within 3 months of Screening.
* History of alcohol abuse or excessive intake of alcohol as judged by the Investigator.
* Positive screen for drugs of abuse, cotinine (nicotine) or alcohol at Screening and/or Day -1.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with myeloperoxidase (MPO) inhibitors and anti-thyroid drugs with similar theorem motifs as AZD4831.
* Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate,) as judged by the Investigator.
* Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega-dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
* Plasma donation within 1 month of Screening or any blood donation/blood loss > 500 mL during the 3 months before Screening.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 1 month of first administration of IMP in this study (period of exclusion begins 1 month after the final dose of the previous chemical entity or last visit in the previous study, whichever is longest),

  1. if the previous chemical entity has a half-life that would not indicate complete clearance at the time of screening to this study,
  2. if the previous chemical entity has significant drug-drug interactions or enzyme inductions that could potentially have an impact on the PK of this study's IMP, even if the previous chemical entity is cleared at the time of screening to this study,
  3. and if the subject has not completed all follow-up activity in the previous study, including last study visit, unresolved AEs, and abnormal laboratory values.
* Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Involvement of any Astra Zeneca, Parexel or study site employee or their close relatives.
* Judgement by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
* Subjects who are vegans or have medical dietary restrictions, or any other dietary restrictions.
* Subjects who cannot communicate reliably with the Investigator.
* Previous bone marrow transplant.
* Non leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male Japanese and Chinese subjects aged 18-50 years
Enrollment: 32 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs)/serious adverse events | Screening through follow-up visit (upto 9 weeks)
  To assess AEs as a variable of safety and tolerability of AZD4831 following oral administration of multiple-ascending doses at steady state in healthy Japanese and Chinese subjects.
Number of subjects with abnormal blood pressure (BP) and pulse | Screening through follow-up visit (upto 9 weeks)
  To assess BP and pulse rate as a variable of safety and tolerability of AZD4831 following oral administration of multiple-ascending doses at steady state in healthy Japanese and Chinese subjects.
Number of subjects with abnormal electrocardiogram (ECG) | Screening through follow-up visit (upto 9 weeks)
  To assess change ECG as a variable of safety and tolerability of AZD4831 following oral administration of multiple-ascending doses at steady state in healthy Japanese and Chinese subjects.
Number of subjects with abnormal abnormal clinical chemistry/hematology/urinalysis | Screening through follow-up visit (upto 9 weeks)
  To assess clinical chemistry/hematology/urinalysis as a variable of safety and tolerability of AZD4831 following oral administration of multiple-ascending doses at steady state in healthy Japanese and Chinese subjects.
Number of subjects with abormal physical examination results | Screening through follow-up visit (upto 9 weeks)
  To assess physical examination as a variable of safety and tolerability of AZD4831 following oral administration of multiple-ascending doses at steady state in healthy Japanese and Chinese subjects.

SECONDARY OUTCOMES:
Plasma Cmax: Maximum observed plasma concentration | Day 1: Pre-dose (pre); 0.25,0.5,1,1.5,2,3,4,6,8,12 h post-dose (post); Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the Cmax of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma Cmax/D | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the Cmax/D of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma tmax: Time to reach peak or maximum observed concentration following drug administration | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the tmax of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma Ctrough: Observed trough plasma concentration | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the Ctrough of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma t1/2λz: Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the t1/2λz of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plamsa AUCτ : Area under the plasma concentration-time curve within the dosing interval | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the AUCτ of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma AUCτ/D | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the AUCτ/D of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma CL/F: Apparent total body clearance of drug from plasma after extravascular administration (Day 10) | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the CL/F of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma Vz/F:Apparent volume of distribution for parent drug at terminal phase after extravascular administration | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the Vz/F of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma AUCinf: Area under the concentration-time curve from time zero extrapolated to infinity | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the AUCinf of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma AUCinf/D: Area under the plasma concentration-time curve from time zero extrapolated to infinity divided by dose | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the AUCinf/D of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma Rac(AUC): Accumulation ratio based upon AUC | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the Rac(AUC) of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Plasma Rac(Cmax): Accumulation ratio based upon Cmax | Day 1: pre; 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 2-9: Pre; Day 10: Pre and at 0.25,0.5,1,1.5,2,3,4,6,8,12 h post; Day 11:24 and 36 h post; Day 12: 48 h post; Day 16:96,144, and 240 h post; Day 24:336 h post
  To characterize the Rac(Cmax) of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Urine Ae(t1-t2): Amount of analyte excreted into the urine from time t1 to t2 | Day1 : Pre; Day 10: 0 to 3, 3 to 6, 6 to 9, 9 to 12, 12 to 24 h post
  To characterize the Ae(t1-t2) of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Urine Ae(0-last): Cumulative amount of analyte excreted at the last sampling interval | Day1 : Pre; Day 10: 0 to 3, 3 to 6, 6 to 9, 9 to 12, 12 to 24 h post
  To characterize the Ae(0-last) of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Urine %fe(t1-t2): Fraction of dose (expressed as a percentage) excreted unchanged into the urine from time t1 to t2 | Day1 : Pre; Day 10: 0 to 3, 3 to 6, 6 to 9, 9 to 12, 12 to 24 h post
  To characterize the %fe(t1-t2) of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Urine %fe(0-last): Percentage of dose excreted unchanged into the urine from time zero to the last measured time point for an analyte | Day1 : Pre; Day 10: 0 to 3, 3 to 6, 6 to 9, 9 to 12, 12 to 24 h post
  To characterize the %fe(0-last) of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.
Urine CLR: Renal clearance of drug from plasma, estimated by dividing Ae(0-last) by AUC(0-t) | Day1 : Pre; Day 10: 0 to 3, 3 to 6, 6 to 9, 9 to 12, 12 to 24 h post
  To characterize the CLR of AZD4831 following multiple-ascending doses in healthy Japanese and Chinese subjects.

CONTACTS AND LOCATIONS:
Overall Officials: David Han, M.D, Principal Investigator — PAREXEL Early Phase Clinical Unit-Los Angeles
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Sunnaker M, Bhattacharya C, Nelander K, Aurell M, Heijer M, Collen A, Han D, Holden J, Trebski M, Garkaviy P, Ericsson H. Pharmacokinetics and Tolerability of the Novel Myeloperoxidase Inhibitor Mitiperstat in Healthy Japanese and Chinese Volunteers. Clin Drug Investig. 2024 Nov;44(11):863-874. doi: 10.1007/s40261-024-01402-x. Epub 2024 Nov 4. PMID 39495467